CLINICAL TRIAL: NCT05695092
Title: Effectiveness of Progressive Muscle Relaxation on Sleep Disturbance in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Waqar Ahmed Awan, Professor, Riphah International University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 01380
Record Dates: First submitted 2023-01-01; First posted 2023-01-23 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Sleep Disturbance in Athletes
MeSH Terms: interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Participant
Masking Description: One group is taking actual intervention and other is taking sham interventioin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): PMR session will be provided a night before competition
  Interventions: Behavioral: Progressive muscle relaxation
- Control group (Sham Comparator): Simple ROM for upper limbs and lower limbs
  Interventions: Other: control

INTERVENTIONS:
Behavioral: Progressive muscle relaxation — Progressive Muscle Relaxation (PMR): This method involved efficiently relaxing global muscles of body with the objective of mental and physical relaxation.
  Other Names: simple Range of Motion
  Arms: Experimental group
Other: control — control group will not receive any intervention
  Arms: Control group

SUMMARY:
Literature supports that athletes have so many reasons for sleep disturbance in their day to day practice and during competition. This study is aimed to build familiarity with the significance of sleep for greatest athletic execution as well as providing Progressoive Muscle Relaxation(PMR),(A technique proposed by Jackobson to improve sleep and degrease the anxiety) as strategy to improve sleep prior to a significant competition during tournament

DETAILED DESCRIPTION:
Adequate sleep is necessary to accomplish ideal athletic performance, cognitive functioning and overall well-being. Inadequate sleep is likewise connected to slow reaction time, delayed perception which can prompt impaired performance and increase risk of injury. A few investigations on sleep and athlete performance have additionally shown that sleep quality can be disturb for so many reasons.

A range of interventions are available that may be beneficial or are commonly utilized in athletes to enhance sleep quantity and quality in athletes. Drug strategies and hypnotics are related with side effects, for example, drug resistance and withdrawal symptoms. Thus, there has been increase in utilization of non-drug strategies for further developing sleep quality. Among such strategies are relaxation methods. It has been considered as one of the cost effective and simple methods for easing sleep. Progressive Muscle Relaxation (PMR) is a method that involved efficiently relaxing global muscles of body with the objective of mental and physical relaxation. PMR is widely used previously to improve sleep in general population however there is currently no evidence to support PMR to improve sleep quality during a competition/tournament as a non-pharmacological method to improve participating athlete's sleep.

The aim of this study is to build familiarity with the significance of sleep for greatest athletic execution as well as providing PMR as strategy to improve sleep prior to a significant competition during tournament.

ELIGIBILITY:
Inclusion Criteria: Participants falling in this category would be recruited into the study.

* Active athletes who are training for a competition.
* Age between 18 -36 years.
* Athletes score falling above 4 on "Athletic Sleep Screening Questionnaire"

Exclusion Criteria:

Participant failing to fall in this category would be excluded of the study.

* Athletes who are not performing for more than a year.
* History of metabolic diseases.
* Athletes taking sleeping aids i.e. sleeping pills.
* Having acute injury

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Sleep quality | Baseline to after 24 hours
  Sleep quality was measured with sleep disturbance score

CONTACTS AND LOCATIONS:
Overall Officials: Professor Waqar Ahmed Awan, PHD, Principal Investigator — FRAHS RIPHAH Islmabad
Locations (1):
- Sports Complex, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No